CLINICAL TRIAL: NCT01310270
Title: The Effects of Omega-3 Fatty Acids Supplementation on Endothelial Function and Inflammation
Acronym: OMEGA-PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-04615
Record Dates: First submitted 2011-03-02; First posted 2011-03-08 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pro-Omega (Experimental): High-dose, short-duration dietary omega-3 fatty acids supplementation
  Interventions: Dietary Supplement: Pro-Omega; Dietary Supplement: Omega 3 Fatty Acid
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Pro-Omega; Dietary Supplement: Omega 3 Fatty Acid

INTERVENTIONS:
Dietary Supplement: Pro-Omega — Pro-Omega, 4.4gm/day x 1 month
Dietary Supplement: Omega 3 Fatty Acid — 4.4 gm/day for 1 month

SUMMARY:
The hypothesis being tested is that in patients with stable claudication and documented PAD, omega-3 supplementation for 1 month will lead to improvement in endothelial function as measured by flow-mediated, brachial artery vasodilation (FMD), as well as improvement in the vascular inflammatory profile as measured by a panel of established circulating inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* intermittent claudication
* resting or exercise Ankle-Brachial Index (ABI) <0.9
* age 50 and more

Exclusion Criteria:

* critical limb ischemia
* hypersensitivity/allergies to fish or seafood
* already on omega-3 fatty acids or equivalent
* significant renal, hepatic, and inflammatory disease
* concurrent severe infections
* acute illness (MI, stroke, major surgery within 30 days)
* receiving immunosuppressive medications or steroids

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | 1 month
  Flow-mediated, brachial artery vasodilation (FMD)

SECONDARY OUTCOMES:
Inflammatory bio-markers | 1 month
  Inflammatory bio-markers: C-reactive protein (hsCRP), interleukin-6 (IL-6), soluble intracellular adhesion molecule-1 (sICAM-1) and the anti-inflammatory mediator 15-epimeric lipoxin

CONTACTS AND LOCATIONS:
Overall Officials: Warren Gasper, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Grenon SM, Owens CD, Nosova EV, Hughes-Fulford M, Alley HF, Chong K, Perez S, Yen PK, Boscardin J, Hellmann J, Spite M, Conte MS. Short-Term, High-Dose Fish Oil Supplementation Increases the Production of Omega-3 Fatty Acid-Derived Mediators in Patients With Peripheral Artery Disease (the OMEGA-PAD I Trial). J Am Heart Assoc. 2015 Aug 21;4(8):e002034. doi: 10.1161/JAHA.115.002034. PMID 26296857
- [Derived] Chong KC, Owens CD, Park M, Alley HF, Boscardin WJ, Conte MS, Gasper WJ, Grenon SM. Relationship between kidney disease and endothelial function in peripheral artery disease. J Vasc Surg. 2014 Dec;60(6):1605-11. doi: 10.1016/j.jvs.2014.08.105. Epub 2014 Oct 16. PMID 25441679
- [Derived] Alley H, Owens CD, Gasper WJ, Grenon SM. Ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery in clinical research. J Vis Exp. 2014 Oct 22;(92):e52070. doi: 10.3791/52070. PMID 25406739
- [Derived] Grenon SM, Owens CD, Alley H, Chong K, Yen PK, Harris W, Hughes-Fulford M, Conte MS. n-3 Polyunsaturated fatty acids supplementation in peripheral artery disease: the OMEGA-PAD trial. Vasc Med. 2013 Oct;18(5):263-74. doi: 10.1177/1358863X13503695. Epub 2013 Sep 19. PMID 24052491